CLINICAL TRIAL: NCT03141359
Title: LCI-LUN-NSC-SBRT-001: Phase II Prospective Trial of Primary Lung Tumor Stereotactic Body Radiation Therapy Followed by Concurrent Mediastinal Chemoradiation and Adjuvant Immunotherapy for Locally-Advanced Non-Small Cell Lung Cancer
Brief Title: Use of High Dose Radiation Followed by Chemotherapy and Radiation to Treat Locally Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081382; 00021247 (Other: Advarra IRB); LCI-LUN-NSC-SBRT-001 (Other: Atrium)
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer Stage II; Lung Cancer Stage III; Non Small Cell Lung Cancer
Keywords: Stereotactic body radiation; Chemoradiation; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Cisplatin; Etoposide; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
  Interventions: Radiation: SBRT; Drug: Carboplatin; Drug: Paclitaxel; Drug: cis Platinum; Drug: Etoposide; Radiation: IMRT; Drug: Durvalumab

INTERVENTIONS:
Radiation: SBRT — Primary tumor SBRT
Drug: Carboplatin — concurrent chemotherapy
Drug: Paclitaxel — concurrent chemotherapy
Drug: cis Platinum — concurrent chemotherapy
Drug: Etoposide — concurrent chemotherapy
Radiation: IMRT — mediastinal radiation
Drug: Durvalumab — adjuvant immunotherapy

SUMMARY:
This is a single-arm, single-stage Phase II study designed to evaluate the 1-year PFS rate in subjects with locally-advanced NSCLC (stage II/III) and treated with Stereotactic Body Radiation Therapy (SBRT) followed by concurrent mediastinal chemoradiation with or without consolidation chemotherapy. A total of 60 subjects will be enrolled to this study over a 4 year accrual period.

DETAILED DESCRIPTION:
This study's primary objective is to assess the efficacy of a treatment regimen involving Stereotactic Body Radiation Therapy (SBRT) delivered to the primary tumor followed by concurrent mediastinal chemoradiation by evaluating the proportion of subjects with locally-advanced non-small cell lung cancer (NSCLC) stage II/III who are alive and progression free at 12 months, and to compare to relevant historical controls. Additionally, the treatment regimen will be evaluated based on progression free survival, overall survival, radiologic clinical complete response rate following completion of therapy, objective response rate as defined by RECIST v 1.1, local and locoregional control, patterns of failure, and quality of life. Safety objectives include the rate of grade 2+ radiation pneumonitis and grade 3+ pulmonary events. Exploratory objectives include differential expression of cytokines and chemokines associated with radiation therapy will be determined.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all the following criteria:

* Histologic or cytologic documentation of NSCLC (all histologies allowed)
* Stage II or III disease (AJCC 7th Edition) based on imaging as required during screening: Stage II disease includes only subjects with medically inoperable N1 disease otherwise meeting eligibility criteria. Primary tumor ≤ 7 cm
* Subjects with non-malignant pleural effusion identified on CT scan are eligible provided the effusion is not known or demonstrated to be an exudative effusion. If a pleural effusion is present, the following criteria must be met to exclude malignant involvement: A pleuracentesis is required if pleural fluid is present and visible on both CT scan and chest x-ray. Pleural fluid cytology must be negative for malignancy. Effusions that are minimal and too small for pleuracentesis as determined by the investigator will be eligible for enrollment.
* FEV1 ≥ 1.0 Liter or ≥ 40% predicted with or without bronchodilator within six months prior to initiation of study treatment. Subjects who meet the criterion without O2, but who need acute (started within 10 days prior to enrollment) supplemental oxygen due to tumor-caused obstruction/hypoxia are eligible, provided the amount of the O2 needed has been stable.
* Age ≥18 years.
* ECOG performance status ≤ 2
* Subjects must have normal organ and marrow function as defined: Leukocytes ≥4,000/mcL; Absolute neutrophil count ≥1,500/mcL; Platelets ≥100,000/mcL; Total bilirubin ≤1.5 times the upper limit of normal; Creatinine clearance ≥25 mL/min/1.73 m2
* Negative serum or urine pregnancy test prior to enrollment for women of childbearing age and potential.
* The effects of radiation on the developing human fetus are not well described. For this reason, women of child-bearing potential and non-sterilized men who are sexually active with a woman of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Must be considered a candidate for durvalumab, per the treating investigator
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

Subjects must not meet any of the following criteria.

* Subjects who have had prior systemic therapy for lung cancer
* Subjects who have had prior radiation to the region of the chest that would result in overlap of radiation therapy fields and determined by the treating physician to impede the treatment of the study malignancy.
* Subjects who are actively being treated on any other interventional research study.
* Prior invasive malignancy unless disease free for a minimum of 3 years from enrollment. However, non-melanoma skin cancer, low risk prostate cancer, well differentiated thyroid cancers, in situ carcinomas of the breast, oral cavity, cervix, and other organs, and tumors that are not thought to impact the life expectancy of the subject according to the treating investigator is permissible.
* Centrally located primary tumor < 2 cm from involved nodal disease which would result in significant overlap of radiation dose. Centrally located is defined as within or touching the zone of the proximal bronchial tree, which is a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus right and left lower lobe bronchi).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2027-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John H Heinzerling, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinzerling JH, Mileham KF, Robinson MM, Symanowski JT, Induru RR, Brouse GM, Corso CD, Prabhu RS, Haggstrom DE, Moeller BJ, Bobo WE, Fasola CE, Thakkar VV, Pal SE, Gregory JM, Norek SL, Begic XJ, Kesarwala AH, Burri SH, Simone CB 2nd. Primary lung tumour stereotactic body radiotherapy followed by concurrent mediastinal chemoradiotherapy and adjuvant immunotherapy for locally advanced non-small-cell lung cancer: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2025 Jan;26(1):85-97. doi: 10.1016/S1470-2045(24)00573-4. Epub 2024 Nov 29. PMID 39615497

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy: SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
  SBRT: Primary tumor stereotactic body radiation therapy (SBRT)
  Concurrent chemotherapy: (Carboplatin + Paclitaxel) or (cis Platinum + Etoposide)
  Mediastinal radiation: intensity-modulated radiation therapy (IMRT)
  Adjuvant immunotherapy: durvalumab
Period: Overall Study
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Started | 61
Completed | 0
Not Completed | 61
Not completed — Death | 32
Not completed — Still On Study (in follow up) | 29

BASELINE CHARACTERISTICS:
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 40
Age, Continuous [Median (Full Range); unit: years] | 67 [50 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 51
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Progression Free and Surviving at 12 Months
Description: 12-month progression free survival was determined for each subject as a binary variable indicating whether or not the subject was progression free and surviving at 12 months after study enrollment. Failure occurred if the subject progressed or died from any cause within 12 months of study enrollment. Disease progression was determined according to RECIST v1.1.
Time Frame: From date of treatment start to date of progression or death, or censored at 12 months, whichever occurred first.
Population: The population evaluable for the 12-month PFS outcome is defined as all subjects who initiate treatment with SBRT and experienced a PFS event within 12 months of enrollment or have at least one year of radiologic follow-up from enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 59
Participants | 37
Statistical Analysis 1: Comparison: SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy; We used a single-stage design to test null hypothesis (H0) that 1-yr PFS is <= 0.60. Assuming one-sided α= 0.10, 60 patients provided 98% power to reject H0, assuming the true 1-yr PFS is 0.80. Since not all enrolled subjects received durva, study power was affected. For patients who did not receive durva, H0 was assumed to be 0.40 versus an alternative of 0.60. Including these subjects reduced power from 98%. The conditional power given that 13 evaluable subjects didn't receive durva was 88%; Test type: Superiority; p = .388, Fisher Exact; Rate = 0.627, 95% CI 2-sided [0.492 to 0.750] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from treatment start date to first occurrence of either progressive disease (PD) or death. PD must be objectively determined per RECIST v1.1 criteria, where progression date is date of last radiologic assessment that identified PD. If subject died without documented PD, progression date will be death date. For surviving subjects who do not have PD, PFS will be censored at the date of last radiologic assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last radiologic assessment prior to commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From date of treatment start to date of progression or death, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted, anticipated posting 2027-07

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from enrollment to the study (treatment start date) to the date of death from any cause. Participants who are alive or lost to follow-up at the time of the analysis will be censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted, anticipated posting 2027-07

4. Secondary Outcome: Radiologic Clinical Complete Response
Description: Radiologic clinical complete response will be recorded for each subject as a binary variable indicating whether or not the subject had no evidence of disease on either PET/CT or CT scan approximately 3 months after the last treatment of concurrent mediastinal chemoradiation.
Time Frame: Approximately 3 months after last treatment of concurrent mediastinal chemoradiation (on average, SBRT plus chemoradiation treatment lasted 2 months from baseline)
Population: Defined as all subjects who initiate treatment with SBRT and who have PET/CT results at approximately 3 months after last treatment of concurrent mediastinal chemoradiation.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 49
Participants | 28
Statistical Analysis 1: Comparison: SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy; Test type: Other — Estimation only; Rate = 0.571, 95% CI 2-sided [0.422 to 0.712] — Confidence interval estimated using the Clopper Pearson method

5. Secondary Outcome: Number of Participants With an Objective Response
Description: Objective response is determined for each participant as a binary variable indicating whether or not the participant achieved a best overall response of complete response (CR) or partial response (PR) as determined by RECIST v1.1 criteria.
Time Frame: From enrollment to best response while on study treatment; participants remained on study treatment (including SBRT, chemoradiation, and durvalumab) 4.5 months on average.
Population: The response evaluable population is defined as all subjects who initiate treatment with SBRT and who have measurable disease present at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 60
Participants | 45
Statistical Analysis 1: Comparison: SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy; Test type: Other — Estimation only; Rate = 0.750, 95% CI 2-sided [0.621 to 0.853] — Confidence interval estimated using the Clopper Pearson method

6. Secondary Outcome: Local Control at 12 and 24 Months
Description: Local control (LC) is defined as the duration of time from enrollment to the study to first progression of the subject's primary lesions(s). If a participant dies prior to local progression local control will be censored at the date of death. For surviving subjects with no documented local progression, local control will be censored at the date of the last radiologic assessment that evaluated the local tumor(s). For subjects who receive subsequent anticancer therapy prior to documented local progression, local control will be censored at the date of last radiologic assessment that evaluated the local tumor(s) prior to the commencement of subsequent therapy. Local control will be estimated at 12 and 24 months.
Time Frame: From date of treatment start to date of progression of primary lesion or censored as described; assessed for approximately 2 years.]
Reporting Status: Not Posted, anticipated posting 2027-07

7. Secondary Outcome: Regional Control at 12 and 24 Months
Description: Regional control (RC) is defined as the duration of time from enrollment to the study to first progression of the subject's regional lesions(s). If a participant dies prior to regional progression regional control will be censored at the date of death. For surviving subjects with no documented regional progression, regional control will be censored at the date of the last radiologic assessment that evaluated the regional tumor(s). For subjects who receive subsequent anticancer therapy prior to documented regional progression, regional control will be censored at the date of last radiologic assessment that evaluated the regional tumor(s) prior to the commencement of subsequent therapy. Regional control will be estimated at 12 and 24 months.
Time Frame: From date of treatment start to date of progression of regional lesions or censored as described; assessed for approximately 2 years.
Reporting Status: Not Posted, anticipated posting 2027-07

8. Secondary Outcome: Locoregional Control at 12 and 24 Months
Description: Locoregional control is defined as the duration of time from enrollment to the study to first progression of the subject's local and/or regional lesions(s), whichever occurs first. If a participant dies prior to locoregional progression locoregional control will be censored at the date of death. For surviving subjects with no documented local and/or regional progression, locoregional control will be censored at the date of the last radiologic assessment that evaluated the local and regional lesion(s). For subjects who receive subsequent anticancer therapy prior to documented locoregional progression, locoregional control will be censored at the date of last radiologic assessment that evaluated the local and regional tumor(s) prior to the commencement of subsequent therapy. Locoregional control will be estimated at 12 and 24 months.
Time Frame: From date of treatment start to date of progression of primary or regional lesions or censored as described; assessed for approximately 2 years.
Reporting Status: Not Posted, anticipated posting 2027-07

9. Secondary Outcome: Distant Control at 12 and 24 Months
Description: Distant control defined as the duration of time from enrollment to first metastatic progression. If a subject dies prior to metastatic progression, distant control will be censored at the date of death. For surviving subjects with no documented metastatic progression, distant control will be censored at the date of the last radiologic assessment. For subjects who receive subsequent anti-cancer therapy prior to documented metastatic progression, distant control will be censored at the date of last radiologic assessment prior to the commencement of subsequent therapy. Distant control will be estimated at 12 and 24 months.
Time Frame: From date of treatment start to date of metastatic progression or censored as described; assessed for approximately 2 years
Reporting Status: Not Posted, anticipated posting 2027-07

10. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Global Health Status Quality of Life Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. EORTC QLQ-C30 includes 5 functional scales, 9 symptom scales/items, and a global health status/quality of life (QoL) scale. The global health status/QoL score is determined from two 7-point items, ranging from 1 (Very Poor) to 7 (Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score represents a higher (better) quality of life.
Time Frame: baseline (pre-SBRT), post-SBRT/pre-chemoradiation, and 1, 3, 6, and 12 months after the last treatment of chemoradiation (on average, SBRT plus chemoradiation treatment lasted 2 months from baseline)
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
score on a scale
  Baseline | 66.25 (2.80)
  Post-SBRT | 62.00 (2.80)
  1 month after Chemoradiation | 65.46 (2.90)
  3 months after Chemoradiation | 64.27 (2.92)
  6 months after Chemoradiation | 64.43 (3.09)
  12 months after Chemoradiation | 60.99 (3.44)

11. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Lung Cancer (EORTC QLQ-LC13) Symptom Scores
Description: The EORTC QLQ-LC13 is a 13-item questionnaire to assess lung cancer associated symptoms, treatment related side effects and pain medication. Both multi-item and single-item measures of lung-cancer associated symptoms and side-effects from conventional chemo and radiotherapy. We focused on 3 symptoms of interest from the EORTC QLQ-LC13: dyspnoea, coughing, and dysphagia. Dyspnoea is a function of three items and can only be determined if all three items have been answered, while coughing and dysphagia are single-item symptoms. Each symptom score is determined by averaging the items that contribute to the scale to get a raw score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher symptom score represents a higher (worse) level of symptoms.
Time Frame: as for outcome 10
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
score on a scale
  Dyspnoea - Baseline | 25.64 (2.97)
  Dyspnoea - Post-SBRT | 26.41 (2.98)
  Dyspnoea - 1 Month After Chemoradiation | 30.91 (3.04)
  Dyspnoea - 3 Month After Chemoradiation | 34.84 (3.06)
  Dyspnoea - 6 Month After Chemoradiation | 31.27 (3.18)
  Dyspnoea - 12 Month After Chemoradiation | 37.28 (3.44)
  Coughing - Baseline | 38.78 (3.41)
  Coughing - Post-SBRT | 38.85 (3.41)
  Coughing - 1 Month After Chemoradiation | 42.86 (3.48)
  Coughing - 3 Month After Chemoradiation | 44.63 (3.53)
  Coughing - 6 Month After Chemoradiation | 44.36 (3.71)
  Coughing - 12 Month After Chemoradiation | 45.29 (4.10)
  Dysphagia - Baseline | 9.37 (2.22)
  Dysphagia - Post-SBRT | 4.56 (2.23)
  Dysphagia - 1 Month After Chemoradiation | 12.38 (2.30)
  Dysphagia - 3 Month After Chemoradiation | 5.24 (2.32)
  Dysphagia - 6 Month After Chemoradiation | 2.48 (2.48)
  Dysphagia - 12 Month After Chemoradiation | 6.19 (2.75)

12. Secondary Outcome: MD Anderson Symptom Inventory - Lung Cancer (MDASI-LC) Total Symptom + Interference Score
Description: The MDASI-LC Module includes 22 questions to assess the severity of multiple lung cancer-related symptoms and the impact of these symptoms on daily functioning. Scores for each item range from 0 to 10, where 0 indicates no symptoms and 10 indicates worst possible symptoms. Arithmetic mean of the items completed was calculated to determine a mean total symptom + interference score ranging from 0 to 10. The mean score is reported if more than 50% of the items are completed on a given administration. Higher scores indicate worse symptoms and more interference.
Time Frame: as for outcome 10
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
score on a scale
  Baseline | 1.56 (0.21)
  Post-SBRT | 1.77 (0.21)
  1 Month After Chemoradiation | 2.05 (0.21)
  3 Months After Chemoradiation | 2.02 (0.22)
  6 Months After Chemoradiation | 1.65 (0.22)
  12 Months After Chemoradiation | 2.34 (0.24)

13. Other Pre Specified Outcome: Number of Participants With Grade 2 or Higher Radiation Pneumonitis
Description: A binary variable will be determined for each subject indicating whether or not the subject experienced at least one grade 2 or higher pneumonitis adverse event according to the NCI Common Terminology for Adverse Events version 4.0 during induction. Pneumonitis events receiving treatment with steroids and possibly, probably, or definitely attributed to SBRT or mediastinal radiation will be included.
Time Frame: From enrollment to 6 months after last treatment of concurrent mediastinal chemoradiation (on average, a total of 8 months).
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 10
Statistical Analysis 1: Comparison: SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy; Test type: Other — Estimation only; Rate = 0.164, 95% CI 2-sided [0.082 to 0.281] — Confidence interval estimated using the Clopper Pearson method

14. Other Pre Specified Outcome: Number of Participants With Grade 3 or Higher Pulmonary Events
Description: A binary variable will be determined for each subject indicating whether or not the subject experienced at least one grade 3 or higher pulmonary adverse event according to the NCI Common Terminology for Adverse Events version 4.0 during induction. This includes pulmonary adverse events regardless of attribution.
Time Frame: Assessed for approximately 12 months after last treatment of concurrent mediastinal chemoradiation (on average, a total of 14 months).
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 15
Statistical Analysis 1: Comparison: SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy; Test type: Other — Estimation only; Rate = 0.246, 95% CI 2-sided [0.145 to 0.373] — Confidence interval estimated using the Clopper Pearson method

15. Other Pre Specified Outcome: Number of Participants With at Least One Serious Event
Description: A binary variable will be determined for each participant indicating whether or not the subject had at least one adverse event that was categorized as serious, regardless of causality. Serious is defined per the study protocol and includes events that the investigator deems serious and results in the following outcomes: death, life-threatening situation, persistent or significant disability/incapacity, requires or prolongs hospitalization, congenital anomaly/birth defect in the offspring of a study participant, suspected transmission of any infections agent via medical product, or based upon medical judgement, may jeopardize the subject and may require medical or surgical intervention to prevent one of the afore listed outcomes from occurring.
Time Frame: as for outcome 14
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 23

16. Other Pre Specified Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event
Description: A binary variable will be determined for each participant indicating whether or not the subject had at least one treatment-emergent adverse event, regardless of causality. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 4.0. Treatment-emergent is defined per the study protocol and includes AEs that occur after treatment start that were not present at the time of treatment start or AEs that increase in severity after treatment start if the event was present at the time of treatment start.
Time Frame: as for outcome 14
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 61

17. Other Pre Specified Outcome: Number of Participants With at Least One Grade 3 or Higher Treatment Emergent Adverse Event
Description: A binary variable will be determined for each participant indicating whether or not the subject had at least one grade 3 or higher treatment-emergent adverse event, regardless of causality. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 4.0. Treatment-emergent is defined per the study protocol and includes AEs that occur after treatment start that were not present at the time of treatment start or AEs that increase in severity after treatment start if the event was present at the time of treatment start.
Time Frame: as for outcome 14
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 41

18. Other Pre Specified Outcome: Number of Participants Who Discontinued Study Treatment Due to Adverse Events
Description: A binary variable will be determined for each participant indicating whether or not the subject discontinued study treatment due to adverse events.
Time Frame: as for outcome 14
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 9

19. Other Pre Specified Outcome: Number of Participants Who Received Durvalumab
Description: A binary variable will be determined for each participant indicating whether or not the subject received at least one dose of durvalumab on study
Time Frame: as for outcome 14
Population: The evaluable population is defined as all subjects who initiate treatment with SBRT.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
Number analyzed (Participants) | 61
Participants | 47

ADVERSE EVENTS:
Time Frame: From enrollment, during treatment, until approximately 12 months after last treatment of concurrent mediastinal chemoradiation (on average, a total of 14 months).
Arm/Group | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy
All-Cause Mortality (participants affected / at risk) | 32/61
Serious Adverse Events (participants affected / at risk) | 23/61
Other Adverse Events (participants affected / at risk) | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy (N=61)
Lung infection (Infections and infestations) | 10
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 — COPD exacerbation
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutrophil count decreased (Investigations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Asthma exacerbation
Acute kidney injury (Renal and urinary disorders) | 1
Bronchial infection (Infections and infestations) | 1
Cardiac disorders - Other (Cardiac disorders) | 1 — CHF exacerbation
Colitis (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Heart failure (Cardiac disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Multi-organ failure (General disorders and administration site conditions) | 1
Sepsis (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT + Concurrent Mediastinal Chemoradiation +/- Consolidation Chemotherapy/Adjuvant Immunotherapy (N=61)
Esophagitis (Gastrointestinal disorders) | 37
Fatigue (General disorders and administration site conditions) | 35
Nausea (Gastrointestinal disorders) | 24
Dysphagia (Gastrointestinal disorders) | 23
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22
Anorexia (Metabolism and nutrition disorders) | 21
Diarrhea (Gastrointestinal disorders) | 21
Constipation (Gastrointestinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16
Non-cardiac chest pain (General disorders and administration site conditions) | 15
Vomiting (Gastrointestinal disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10
Lung infection (Infections and infestations) | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 9
Edema limbs (General disorders and administration site conditions) | 9
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 9
Chest wall pain (Musculoskeletal and connective tissue disorders) | 8
Dysgeusia (Nervous system disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 7
Dizziness (Nervous system disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hypothyroidism (Endocrine disorders) | 7
Pain (General disorders and administration site conditions) | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Sinus tachycardia (Cardiac disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Anemia (Blood and lymphatic system disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Hypotension (Vascular disorders) | 5
Mucosal infection (Infections and infestations) | 5
Paresthesia (Nervous system disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 — COPD exacerbation
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 — hemoptysis
Skin infection (Infections and infestations) | 5
Upper respiratory infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5
White blood cell decreased (Investigations) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Infusion related reaction (General disorders and administration site conditions) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Weight loss (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT03141359/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT03141359/ICF_000.pdf